CLINICAL TRIAL: NCT04746469
Title: Impact of Automated Telephone Outreach on Colorectal Cancer Screening Uptake Among Patients Who Receive Mailed Fecal Immunochemical Tests (FIT)
Brief Title: Using Behavioral Science to Improve Colorectal Cancer Screening Rates With Mailed FIT Kits
Acronym: FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel M. Croymans, MD, MBA, MS, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB #19-001418
Record Dates: First submitted 2021-01-24; First posted 2021-02-09 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer Screening

STUDY DESIGN:
Intervention Model Description: ~2500 patients who are overdue for average-risk CRC screening and are enrolled in UCLA Health biannual mailed FIT program will be randomized to either control (mailed FIT kit + standard messaging) or intervention (mailed FIT Kit + standard messaging + delayed automated phone reminder)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group will receive standard FIT mailer protocol (includes mailed FIT kit plus standardized messaging via EHR portal)
- Intervention (Experimental): This group will receive standard FIT mailer protocol (as above) PLUS delayed automated phone reminder
  Interventions: Behavioral: Delayed automated phone call

INTERVENTIONS:
Behavioral: Delayed automated phone call — Cipher provides automated phone calls to patients; in this case the script for Cipher was modified to provide patients a reminder to return FIT kits, allow patients to request a new kit in case they need a replacement, and to allow patients to provide information if they already completed CRC screening
  Other Names: Cipher phone reminder
  Arms: Intervention

SUMMARY:
As a part of UCLA Health's continued goal of improving patient care the investigators are updating our mailing campaign for our FIT Kit colorectal cancer screening that the investigators administer 2 times per year to include an automated phone call reminder to patients who are overdue for average-risk colorectal cancer screening and enrolled in a mailed FIT program. This will help the investigators evaluate if automated phone calls are effective at improving compliance with CRC screening, in addition to mailed FIT and embedded electronic health record (EHR) portal messages to patients.

DETAILED DESCRIPTION:
UCLA Health has a biannual mailed FIT program designed to capture patients overdue for CRC screening who are average-risk for CRC. With every campaign, the investigators attempt to improve the return rates for patients receiving the FIT Kits. For the current campaign, all patients enrolled will receive usual care and the investigators are delivering an automated phone call to half the eligible patients reminding them to return their FIT kits and prompting them to request a new kit if needed. The investigators will investigate if this intervention increases the number of patients who complete the mailed Fit Kit or any type of CRC screening over a 6-month follow up period. This quality improvement project will help the investigators improve the processes of care for the patients, and community. If this phone call is successful the investigators will likely expand it to the entire population in future FIT Kit mailer campaigns. However, if it is not effective this will help the investigators minimize the number of calls/interventions the investigators send to patients and will hopefully allow for more useful outreach to patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Overdue for average-risk colorectal cancer screening
* Active primary care provider at UCLA seen within last 3 years

Exclusion Criteria:

* Inactive mychart status at time of enrollment
* Died within follow-up period
* Received FIT kit in prior 6 months

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Overall colorectal cancer screening uptake (any modality) | 6 months
  Rate of completion of CRC screening by any of the following: FIT, colonoscopy, CT colonography, sigmoidoscopy or FIT-DNA within study period.

SECONDARY OUTCOMES:
Colorectal cancer screening uptake by modality | 6 months
  Rate of completion of CRC screening by modality type

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Health Department of Medicine, Quality Office, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No